CLINICAL TRIAL: NCT05018208
Title: Remote Monitoring in Cancer Care: A Platform Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC211001; NCI-2021-07955 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-002043 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-08-03; First posted 2021-08-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma; Hematopoietic and Lymphoid Cell Neoplasm; Lung Carcinoma; Malignant Digestive System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms | interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Arm 1 (wearable device[s], smartphone app): Patients undergoing CAR-T therapy use the Biofourmis wearable device(s) and smartphone app to answer a series of questions about health and neurologic symptoms a few times a day for 5 weeks.
  Interventions: Other: Computer-Assisted Intervention; Procedure: Patient Monitoring
- Arm 2 (wearable device[s], smartphone app, questionnaires): Patients undergoing radiation therapy (RT) for head and neck, lung, or gastrointestinal cancers use the Biofourmis wearable device(s) for 90 days after completion of RT. Patients also use the smartphone app to answer a series of questions about health and neurologic symptoms before start of RT, after completion of RT, 3 months after completion of RT, and 1 year after completion of RT. In addition, patients complete weekly questionnaires regarding side effects and tolerance of the device.
  Interventions: Other: Computer-Assisted Intervention; Procedure: Patient Monitoring; Other: Questionnaire Administration

INTERVENTIONS:
Other: Computer-Assisted Intervention — Use smartphone app
Procedure: Patient Monitoring — Wear Biofourmis wearable device(s)
  Other Names: medical monitoring; monitor
Other: Questionnaire Administration — Complete questionnaires
  Groups: Arm 2 (wearable device[s], smartphone app, questionnaires)

SUMMARY:
This study investigates a device that closely monitors vital signs, as well as a smartphone application (app) that allows patients to respond to different questions and tests that will monitor for new symptoms. This study may help researchers understand if wearing the device is a better tool than standard vital sign assessment tools done only while at the doctor's office or hospital, and if using the smartphone app is a better tool than standard assessment tools used while in the doctor's office or hospital.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop patient-specific algorithms to predict the trajectory of cytokine release syndrome (CRS) and or neurotoxicity and time to escalation of medical intervention is needed. (Arm 1) II. Establish the validity for the use of mobile technology to assess neurologic symptoms remotely. (Arm 1) III. Compare the time to escalation of potential medical intervention between remote monitoring (RM) and standard care (SC) based on retrospective analysis of clinical trial data. (Arm 1) IV. Establish the feasibility for the use of wearable device for continuous, remote monitoring of physiologic parameters by quantifying false alerts and downstream clinical actions. (Arm 1) V. Define the range of physiologic variables associated with receipt of radiation and chemotherapy. (Arm 2) VI. Correlate PROs and physician rated CTCAE to biologic parameters. (Arm 2) VII. Establish the feasibility for the use of wearable device for continuous, remote monitoring of physiologic parameters by quantifying false alerts and downstream clinical actions. (Arm 2)

OUTLINE:

ARM 1: Patients undergoing CAR-T therapy use the Biofourmis wearable device(s) and smartphone app to answer a series of questions about health and neurologic symptoms a few times a day for 5 weeks.

ARM 2: Patients undergoing radiation therapy (RT) for head and neck, lung, or gastrointestinal cancers use the Biofourmis wearable device(s) for 60 to 90 days after completion of RT. Patients also use the smartphone app to answer a series of questions about health and neurologic symptoms before start of RT, after completion of RT, 3 months after completion of RT, and 1 year after completion of RT. In addition, patients complete weekly questionnaires regarding side effects and tolerance of the device.

ELIGIBILITY:
Inclusion Criteria:

* ARM 1: Age >= 18 years
* ARM 1: Provide written informed consent
* ARM 1: Patients undergoing commercial CAR-T cell therapy in an outpatient setting
* ARM 2: Age >= 18 years
* ARM 2: Provide written informed consent
* ARM 2: Patients with a plan to undergo radiation therapy for lung, gastrointestinal, or head and neck cancer

Exclusion Criteria:

* ARM 1: Non-English speaking
* ARM 1: Planned initiation of lymphodepleting chemotherapy in the inpatient setting
* ARM 2: Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing standard of care CAR-T cell therapy in the outpatient setting at Mayo Clinic. Patients undergoing standard of care radiation for (1) head and neck, (2) lung, or (3) gastrointestinal malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of remote monitoring-based CRS detection/ prediction (Arm 1) | Up to 5 weeks
Assessment of neurotoxicity via digital capture of neurological assessment (Arm 1) | Up to 5 weeks
  Will assess agreement and concordance between assessment of neurotoxicity via digital capture of neurological assessment (ICE) as compared to standard in-person assessment.
BF-Mayo Neuro test (Arm 1) | Up to 5 weeks
  Will assess agreement and concordance between BF-Mayo Neuro test and ICE-based assessment of neurotoxicity.
Sensitivity, specificity, positive predictive value and negative predictive value of novel digital neurotoxicity tests (BF-Neuro) (Arm 1) | Up to 5 weeks
  Will compare to standard in-person ICE based neurotoxicity assessment.
Range of physiologic variables associated with receipt of radiation and chemotherapy (Arm 2) | Up to 1 year
Quantification of false alerts and downstream clinical actions (Arm 2) | Up to 1 year
  Will be used for the establishment of the feasibility for the use of wearable device for continuous, remote monitoring of physiologic parameters.

SECONDARY OUTCOMES:
Biovital index (Arm 1) | Up to 5 weeks
  Will assess correlation between Biovital index and BF-Mayo Neuro Test and adverse clinical events. Both continuous variables (physiologic parameters) and categorical variables (events) will be used to generate a mixed effects logistic regression model with repeated measures. The goal is to identify patterns of changes in the continuous data associated with either clinically relevant or significant events.
BF-Mayo Neuro Test (Arm 1) | Up to 5 weeks
  Will assess correlation between Biovital index and BF-Mayo Neuro Test and adverse clinical events. Both continuous variables (physiologic parameters) and categorical variables (events) will be used to generate a mixed effects logistic regression model with repeated measures. The goal is to identify patterns of changes in the continuous data associated with either clinically relevant or significant events.
Point-in-time assessment of physiological signals from wearable devices (Arm 1) | Up to 5 weeks
  Will assess agreement and concordance from wearable vs. standard of care devices. Intraclass correlation coefficients (ICC) and Bland-Altman methods will be used for agreement and concordance analysis of the remote monitor reading compared to the "gold standard" standard of care devices.
Point-in-time assessment of physiological signals from standard of care devices (Arm 1) | Up to 5 weeks
  Will assess agreement and concordance from wearable vs. standard of care devices. ICC and Bland-Altman methods will be used for agreement and concordance analysis of the remote monitor reading compared to the "gold standard" standard of care devices.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Paludo, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials